CLINICAL TRIAL: NCT05113017
Title: To Evaluate the Effectiveness and Safety of Stereotactic Radiotherapy (SBRT) in the Treatment of Patients With Residual Malignant Pulmonary Nodules After Lung Cancer Surgery: A Multi-center, Prospective Clinical Trial (SMILE)
Brief Title: The Effectiveness and Safety of SBRT in the Treatment of Patients With MPLC After Surgery (SMILE)
Acronym: SMILE
Status: Recruiting | Type: Observational
Sponsor: Fang Wu (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Hunan Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Fang Wu, Clinical Associate Professor, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Other Study IDs: XYEYY20210728
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: The Efficacy and Safety of SBRT in MPLC
Keywords: SBRT, MPLC, Efficacy, Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBRT group: Patients with residual lung nodules are treated with SBRT
  Interventions: Other: NO Intervention

INTERVENTIONS:
Other: NO Intervention — NO Intervention

SUMMARY:
To prospectively evaluate the effectiveness and safety of SBRT in the treatment of residual malignant pulmonary nodules after lung cancer, and is committed to providing new treatment options for patients with multiple primary malignant pulmonary nodules who cannot tolerate multiple operations.

ELIGIBILITY:
Inclusion Criteria:

(1) Age 18-75 years old; (2) ECOG score 0-2 points; (3) Chest CT showed at least two lung nodules (pure ground glass, partial solid or solid nodules); (4) At least one lesion has been pathologically diagnosed as lung cancer (T1N0M0-T1N1M0); (5) At least one residual pulmonary nodule has been diagnosed pathologically or multidisciplinary diagnosis and treatment (MDT) discussed and considered as a primary malignant pulmonary nodule; (6) The residual lung nodules are inoperable or operable but the patient refuses to be surgically removed; (7) Have self-consciousness and can sign informed consent; (8) Must be able to swallow tablets.

Exclusion Criteria:

(1) There are metastatic pulmonary nodules; (2) Have received chest radiotherapy in the past; (3) Lymph node metastasis or distant metastasis; (4) The tumor is located in the proximal bronchial tree area. The proximal bronchial tree is defined as carina, left and right main bronchus, left and right upper lobe bronchus, middle bronchus, right middle lobe bronchus, lingual bronchus, left and right lower lobe bronchi; the proximal bronchial tree area is defined as surrounding the proximal bronchial tree in all directions The area within 2cm above; (5) Pneumonectomy patients; (6) Severe primary diseases such as heart, liver, kidney, hematopoietic system, etc.; (7) Women during pregnancy and lactation; (8) Active period of the human immunodeficiency virus (HIV) infection; (9) Those with active systemic infection, pneumonia, tuberculosis, and pericarditis; (10) There is a history of psychotropic drug abuse or drug abuse;(11)Insulin dependent diabetes;(12) Thyroid disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable residual malignant nodules after early multiple primary lung cancer surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local control rate of cancer of SBRT | 2-year
  Local control rate of cancer
Incidence of Treatment-Emergent Adverse Events of SBRT [Safety and Tolerability] | 2-year
  Treatment-related adverse event

SECONDARY OUTCOMES:
Survival | 2-year
  Survival rate without local recurrence
Survival | 2-year
  Survival rate without distant metastasis
PFS | 2-year
  Progression-free survival rate
OS | 2-year
  Overall survival rate

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Oncology Department，Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha
  - The Third Xiangya Hospital, Central South University, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided